CLINICAL TRIAL: NCT01764243
Title: A Double-Blind, Placebo-Controlled Phase2 Study of MT-4666 in Patients With Mild to Moderate Probable Alzheimer's Disease.
Brief Title: Safety and Efficacy of MT-4666
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P211-03
Record Dates: First submitted 2012-12-26; First posted 2013-01-09 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Nicotinic Acetylcholine Receptor Agonist; Cognitive function; Dementia; Central Nervous System Agents
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- MT-4666 Low Dose (Experimental): low dose
  Interventions: Drug: MT-4666
- MT-4666 High Dose (Experimental): high dose
  Interventions: Drug: MT-4666
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT-4666 — low dose, high dose
  Arms: MT-4666 High Dose; MT-4666 Low Dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the safety and efficacy as assessed by the Alzheimers Disease Assessment Scale-cognitive subscale 13-item (ADAS-cog-13) of two doses of MT-4666 or placebo administered daily for 24 weeks to subjects with mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Probable Alzheimer's disease consistent with National Institute of Neurological and Communicative Disorders and Stroke (NINCDS) and Alzheimer's Disease and Related Disorders Association (ADRDA) criteria
* MMSE score of 10 to 24 inclusive at screening and at Day 1, and CDR-SB score of ≥ 2 at screening
* Modified Hachinski Ischemic Score (mHIS) ≤ 4 at screening
* Caregiver available; caregiver sees subject at least four days (at least 12 hours) each week
* Subject living at home; if living at senior residential setting, or an institutional setting, subject with caregiver indicated above is available

Exclusion Criteria:

* Inability to perform cognitive tests (ADAS-cog-13 and MMSE) at screening and at Day 1
* Diagnosis of any other disease which may cause dementia
* MRI or CT scan within 6 months before screening, with findings inconsistent with the diagnosis of Probable AD
* Diagnosis of major depressive disorder as defined by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) within last five years
* History of or current diagnosis of any psychosis
* History of myocardial infarction or unstable angina within six months before screening
* History of cerebrovascular disorder within 18 months before screening

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2012-11; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in ADAS-cog-13 | Baseline and Week 24

SECONDARY OUTCOMES:
Change from baseline in Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) | Baseline and Week 24
Change from baseline in Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) | Baseline and Week 24
Change from baseline in Alzheimers Disease Assessment Scale-cognitive subscale 11-item (ADAS-cog-11) | Baseline and Week 24
Change from baseline in Mini-Mental State Examination (MMSE) | Baseline and Week 24
Change from baseline in Neuropsychiatric Inventory (NPI) | Baseline and Week 24
Change from baseline in Modified Crichton Scale | Baseline and Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Yu Nakamura, M.D., Ph.D., Study Director — Kagawa University School of Medicine; Akira Homma, M.D., Study Director — Tokyo Dementia Care Research and Training Center; Shun Shimohama, M.D., D. Med. SC, Study Director — Sapporo Medical University
Locations (1):
- Kanto, Japan